CLINICAL TRIAL: NCT01592084
Title: Cohort Study of the Relationship of Hyperlipidemia and Statin Therapy on Survival and Disease Progresssion in Amyotrophic Lateral Sclerosis
Brief Title: Hyperlipidemia and Statin Therapy in Amyotrophic Lateral Sclerosis
Status: Completed | Type: Observational
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Sharon Halton, Research Coordinator, The Methodist Hospital Research Institute
Other Study IDs: IRB(2)0609-0087
Record Dates: First submitted 2012-04-13; First posted 2012-05-07 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: lipid lowering therapy; survival; ALSFRS; age; BMI; weight
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Body Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- lipid lowering therapy: those with lipid lowering therapy those without lipid lowering therapy

SUMMARY:
The role of hyperlipidemia and lipid lowering therapy (LLT) in Amyotrophic Lateral Sclerosis (ALS) pathophysiology and its impact on disease progression and survival is unclear. The investigators analyzed the correlation between lipid levels with disease progression and survival in ALS patients and the association of LLT with these outcomes.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of laboratory-supported probable, probable, or definite familial, sporadic ALS, according to a modified El Escorial criteria (ref), by the study investigators
* Time from disease onset is less than three years

  * 18 years of age
* Subjects with diagnosis of hyperlipidemia and/or taking lipid lowering medications will not be excluded from study.

Exclusion Criteria:

* Requirement for tracheotomy ventilation or non-invasive ventilation for > 23 hours per day
* Diagnosis of other neurodegenerative diseases (Parkinson disease, Alzheimer disease, etc)
* A clinically significant history of significant medical illness (advanced cancer, chronic inflammatory/infectious conditions, etc) within six months of baseline
* Use of progestins, anabolic steroids, and corticosteroids within 45 days of baseline visit. Therapy is allowed as medically indicated after baseline visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the Methodist Neurological Institute
Sampling Method: Probability Sample
Enrollment: 267 (Actual)
Dates: Start 2008-04; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
survial(tracheostomy free,<23 hours on NIPPV, from enrollment) | 3years
  Death was confirmed from Social Security Death Index or newspaper obituaries. Tracheostomy- ventilation was also considered as an end of the life time point.

SECONDARY OUTCOMES:
ALSFRS(measure of disability) | at first evaluation(time 0-T0) to six months (T6)
  DeltaFS = (48-ALSFRS at first evaluation )/duration from onset to diagnosis (month) changeFS=(ALSFRS at six months-ALSFRS at first evaluation)/6

CONTACTS AND LOCATIONS:
Overall Officials: Ericka P Simpson, M.D, Study Director — the Methodist Neurological Institute
Locations (1):
- the Methodist Neurological Institute, Houston, Texas, United States